CLINICAL TRIAL: NCT05052931
Title: Nab-paclitaxel Combined With Oxaliplatin and S-1 for Perioperative Treatment of Advanced Gastric Cancer, a Small-scale, Exploratory Real-world Study
Brief Title: Nab-paclitaxel Combined With Oxaliplatin and S-1 for Perioperative Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianjun Yang (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jianjun Yang, Director, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KIL-GC-006
Record Dates: First submitted 2021-08-25; First posted 2021-09-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Nab-paclitaxel combined with oxaliplatin and S-1
  Interventions: Drug: Nab-paclitaxel combined with oxaliplatin and S-1

INTERVENTIONS:
Drug: Nab-paclitaxel combined with oxaliplatin and S-1 — Nab-paclitaxel 100mg/m^2, D1, Q3W; oxaliplatin 85 mg/m^2, D1, Q3W; S-1 60 mg/m^2, D1-14, Q3W; Neoadjuvant chemotherapy 2 cycles, followed by surgery, continue to receive 6 cycles of adjuvant chemotherapy.

SUMMARY:
This is a prospective, single-center, open, historically controlled real-world study.

The aims of this study is to evaluate the safety and effectiveness of Nab-paclitaxel combined with oxaliplatin and S-1 in the treatment of patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma diagnosed by histology.
* Ambulatory cases, 18-75 years old
* ECOG performance status ≤ 1
* Have not received anti-tumor therapy previously (such as surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy)
* Patients able to tolerate abdominal surgery above grade 3
* Has adequate organ function as defined by the following criteria:

  * WBC> 4.0×10^9/L
  * ANC> 1.5×10^9/L
  * ANC ≥ 1.5×10^9/L
  * HB ≥ 80 g/L
  * PLT ≥ 100×10^9/L
  * TBIL ≤ 1.5×ULN
  * ALT and AST <2.5 × ULN, for patients with liver metastases, ALT and AST <5 × ULN
  * BUN and Cr ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 50 mL/min
* No history of other tumors
* Be willing and able to comply with the plan during the research period
* Has given written informed consent
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Those with a history of other malignancies in the last 5 years, except for cured non-melanoma skin cancer and cervical carcinoma in situ
* HER-2+ and willing to receive Trastuzumab
* Pregnancy or breast-feeding women; Men and women who are sexually active (possible to have children) and unwilling to use contraception during the study period
* Severe, uncontrolled medical diseases and infections; chronic bowel disease or short bowel syndrome
* Major organ failure, such as compensatory cardiopulmonary liver and kidney failure; severe liver and kidney metabolism abnormalities, affecting the normal metabolism of drugs
* Patients with other surgical contraindications, such as serious diseases that are difficult to control
* The researcher believes that patients with a clear gastrointestinal bleeding tendency and/or patients with abnormal blood coagulation function (INR > 1.5)
* Active HBV or HCV
* Peripheral neuropathy ≥ Grade 2 according to NCT-CTC AE5.0
* Patients who are allergic to the drugs in this study, or determined by the investigator as unsuitable to participate in this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
AE | 2-year
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE V5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | 7-month
  ORR is defined as the rate of complete response (CR) or partial response (PR), as determined by IRC using RECIST v1.1 criteria among patients with at least one target lesion.
Disease Control Rate (DCR) | 7-month
  The proportion of all subjects who assessed the best overall curative effect as CR, PR, and disease stable (SD) according to the RECIST 1.1 standard.
Overall survival (OS) | 2-year
  It is defined as the time from the first doses durg to the time of death due to any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi'an, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng J, Wang S, Xu G, Wang J, Wang Y, Luo J, Wang Y, Yang J. A small-scale, exploratory real-world study of nab-paclitaxel combined with oxaliplatin and tegafur in the perioperative treatment of advanced gastric cancer: a study protocol for a real-world clinical trial. J Gastrointest Oncol. 2023 Apr 29;14(2):1131-1140. doi: 10.21037/jgo-23-131. Epub 2023 Apr 27. PMID 37201078